CLINICAL TRIAL: NCT07244705
Title: An Open-label, Multicenter, Phase 1/2 Study Exploring the Safety and Efficacy of ABT-301 in Combination With Tislelizumab and Bevacizumab in Participants With Proficient Mismatch Repair (pMMR)/Non-Microsatellite Instability-High (Non-MSI-H) Locally Advanced or Metastatic Colorectal Cancer (mCRC)
Brief Title: A Study of ABT-301 Plus Tislelizumab With Bevacizumab in pMMR/Non-MSI-H Locally Advanced or mCRC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anbogen Therapeutics, Inc. (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABT-301-103
Record Dates: First submitted 2025-11-10; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer (Diagnosis); Colorectal Cancer Metastatic; Colorectal Cancer (CRC); Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Disease | interventions — 3-(1-benzenesulfonyl-2,3-dihydro-1H-indol-5-yl)-N-hydroxyacrylamide; tislelizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Dose Escalation Phase) (Experimental)
  Interventions: Drug: ABT-301; Drug: Tislelizumab; Drug: Bevacizumab (Avastin)
- Part 2 (Dose Optimization Phase) (Experimental)
  Interventions: Drug: ABT-301; Drug: Tislelizumab; Drug: Bevacizumab (Avastin)

INTERVENTIONS:
Drug: ABT-301 — ABT-301 is an oral histone deacetylase inhibitor (HDACi) administered in capsule form once daily (QD ±3 hours) or every 12 hours (Q12H ±3 hours, with at least 9 hours between doses) with water in 21-day treatment cycles.
  In Part 1 (dose-escalation phase), participants receive escalating doses of ABT-301 (50 mg QD, 100 mg QD, 50 mg Q12H, 150 mg QD, or 75 mg Q12H). Tislelizumab 200 mg and bevacizumab 7.5 mg/kg will be administered through IV infusion on Day 1 of every 21-day treatment cycle. This phase aims to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of ABT-301 when combined with tislelizumab and bevacizumab.
  In Part 2 (dose-optimization phase), two ABT-301 doses/schedules will be selected for further evaluation of antitumor activity, safety, and tolerability in adults with pMMR/non-MSI-H colorectal cancer (CRC).
  Other Names: MPT0E028; Imofinostat
Drug: Tislelizumab — Tislelizumab is a humanized immunoglobulin G4-variant monoclonal antibody (mAb) blocking programmed cell death protein 1 (PD-1). Tislelizumab 200 mg will be administered through IV infusion on Day 1 of every 21-day treatment cycle in combination with ABT-301 and bevacizumab throughout both parts of the study.
Drug: Bevacizumab (Avastin) — Bevacizumab (Avastin®) is a recombinant humanized monoclonal IgG1 antibody which binds to and neutralizes VEGF. Neutralization of VEGF by bevacizumab has been shown to inhibit the VEGF-induced proliferation of human endothelial cells in vitro and to decrease micro-vessel density and interstitial pressure in tumor xenografts in vivo. Bevacizumab 7.5 mg/kg will be administered through IV infusion on Day 1 of every 21-day treatment cycle in combination with ABT-301 and tislelizumab, throughout both parts of the study.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of escalating doses of ABT-301 in combination with fixed doses of tislelizumab 200 mg IV infusion and bevacizumab 7.5 mg/kg IV infusion Q3W, in participants with pMMR/non-MSI-H colorectal cancer (CRC). It will also determine the maximum tolerated dose (MTD) and select the recommended Phase 2 dose (RP2D) of ABT-301.

Participants will receive ABT-301 administered once daily (QD ±3 hours) or twice daily (Q12H ±3 hours, at least 9 hours apart) with water in 21-day treatment cycles. Tislelizumab 200 mg IV and bevacizumab 7.5 mg/kg IV Q3W will be given in both parts of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 years at the time of signing the informed consent.
* Participant with pMMR/non-MSI-H advanced/recurrent histologically confirmed CRC with at least one measurable lesion, per RECIST version 1.1.
* Participant must have received ≥2 lines of prior systemic therapy (including but not limited to chemotherapeutic agents of 5-fluorouracil, oxaliplatin, irinotecan; participant may or may not have received biologic agents such as cetuximab, panitumumab, aflibercept, ramucirumab, bevacizumab; tyrosine kinase inhibitors of regorafenib, fruquintinib).

NOTE: Participants with BRAF V600E, HER2 amplification/ mutation, KRAS G12C mutation, NTRK gene fusion, RET fusion, may or may not have received relevant targeted therapy and failed.

* Participant must submit an archival formalin-fixed, paraffin-embedded tumor specimen collected within 5 years before screening. If archival specimens are unavailable, alternative samples, such as colon endoscopy biopsy, are acceptable.

NOTE: For participants who consent to join the exploratory biomarker study, a fresh biopsy sample is required during the screening and treatment periods. Exceptions may be granted if tumor tissue cannot be obtained due to specific circumstances.

* Tumor tissues were identified as pMMR by immunohistochemistry (IHC) method or nonMSI-H by polymerase chain reaction (PCR) (Appendix 13).
* ECOG Performance Status of 0 or 1.
* Adequate hematologic and end-organ function, defined by laboratory data obtained within 7 days prior to the first dose of study intervention:

  1. Absolute neutrophil count ≥1.5 × 109/L (1500/μL) without granulocyte colony-stimulating factor support.
  2. Lymphocyte count >0.5 × 109/L (500/µL).
  3. Platelet count >100 × 109/L (100,000/μL), without transfusion.
  4. Hemoglobin >90 g/L (9 g/dL), participants may be transfused to meet this criterion.
  5. AST, ALT, and ALP <2.5 × ULN (must be ≤5 × ULN for participants with liver metastases).
  6. Total serum bilirubin <1.5 × ULN (<3 × ULN in the presence of documented Gilbert's syndrome [unconjugated hyperbilirubinemia] or liver metastases at baseline).
  7. Creatinine clearance >60 mL/min.
  8. Serum albumin ≥30 g/L (3 g/dL).
  9. International normalized ratio (INR) or activated partial thromboplastic time (aPTT) <1.5 × ULN.
  10. Urine dipstick for proteinuria ≤2+ (within seven days prior to the first dose of study intervention).
* Resolution of any acute, clinically significant treatment-related toxicity from prior therapy to Grade ≤1 prior to study entry, with the exception of Grade ≤2 chemotherapy-related peripheral neuropathy or any Grade alopecia.
* Participant must have a negative test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, or human immunodeficiency virus (HIV) antibody.

NOTE: Participants with active hepatitis B virus (HBV) infection are eligible for the study if the following applies: HBV deoxyribonucleic acid (DNA) <500 IU/mL within 28 days prior to initiation of study intervention, and anti-HBV treatment (per local standard of care, e.g., entecavir) for a minimum of 14 days prior to study entry and willingness to continue treatment for the length of the study. Participants with positive hepatitis C virus (HCV) test are eligible for the study if they complete their antiviral therapy prior to study entry.

* Contraceptive use by participants or participant partners must be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

NOTE: The reliability of sexual abstinence for male and/or female enrollment eligibility needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post ovulation methods) and withdrawal are not acceptable methods of contraception.

Male Participants:

A male participant must agree to use a highly effective contraception as detailed in Appendix 4 of this protocol during the intervention period and for at least 90 days after the last dose of study intervention and refrain from donating sperm during this period.

Female Participants:

A female participant is eligible to participate if she is not pregnant (see Appendix 4), not breastfeeding, and at least one of the following conditions applies:

o Not a CBP participant as defined in Appendix 4 and below: surgically sterile (documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy as confirmed by review of the participant's medical records, medical examination, or medical history interview), or postmenopausal (defined as no menses for 12 months) without an alternative medical cause with follicle-stimulating hormone (FSH) level in the postmenopausal range ≥1 year.

OR

o A CBP participant who agrees to follow the contraceptive guidance in Appendix 4 during the intervention period and for at least 180 days after the last dose of study intervention.

- Participant is capable of giving signed informed consent as described in Appendix 1, Section 10.1.3 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* History of leptomeningeal disease.
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, psoriatic arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis, or ankylosing spondylitis.

EXCEPTIONS:

* Participants with the following conditions are eligible for the study: autoimmune-related hypothyroidism on thyroid-replacement hormone are eligible for the study. Participants with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
* Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., participants with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met: 1. Rash must cover <10% of body surface area 2. Disease is well controlled at baseline and requires only low-potency topical corticosteroids 3. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.

  * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.

EXCEPTIONS:

o History of radiation pneumonitis in the radiation field (fibrosis) is permitted.

* Active tuberculosis.
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within three months prior to initiation of study intervention, unstable arrhythmia, or unstable angina.

NOTE: Participants are not eligible for the study if they have or are

1. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds).
2. A history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
3. Using concomitant medications that prolong the QT/QTc interval. - Major surgical procedure, other than for diagnosis, within four weeks prior to initiation of study intervention, or anticipation of need for a major surgical procedure during the study.

   * History of malignancy other than CRC within five years prior to screening.

   EXCEPTIONS:

   o Participants with malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer, are eligible for the study.

   - Severe infection within four weeks prior to initiation of study intervention, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.

   - Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the participant at high risk from treatment complications.

   - History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
   * Known hypersensitivity to Chinese hamster ovary cell products or to any component of the tislelizumab or bevacizumab formulation.
   * Participant is breastfeeding, has a positive serum pregnancy test at the Screening Visit, or is planning to become pregnant during the study intervention or within at least 120 days after the last dose of study intervention.
   * Symptomatic, untreated, or actively progressing CNS metastases.

   NOTE: Asymptomatic participants with treated CNS lesions are eligible, provided that all of the following criteria are met:
   * Measurable disease, per RECIST version 1.1.
   * Must be present outside the CNS.
   * The participant has no history of intracranial hemorrhage or spinal cord hemorrhage.
   * There is no evidence of interim progression between completion of CNS-directed therapy and initiation of study intervention.
   * The participant has not undergone stereotactic radiotherapy within seven days prior to initiation of study intervention, whole brain radiotherapy within 14 days prior to initiation of study intervention, neurosurgical resection within 28 days prior to initiation of study intervention.
   * The participant has no ongoing requirement for corticosteroids as therapy for CNS disease.

   NOTE: Anticonvulsant therapy at a stable dose is permitted. Asymptomatic participants with CNS metastases newly detected at screening are eligible for the study after receiving radiotherapy or surgery, with no need to repeat the screening brain scan.
   * Uncontrolled tumor-related pain:

<!-- -->

1. Participants requiring pain medication must be on a stable regimen at study entry.
2. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Participants should recover from the effects of radiation. There is no required minimum recovery period.
3. Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.

   * Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).
   * Treatment with any investigational therapy within 28 days prior to initiation of study intervention.
   * Treatment with the following pharmaceutical or herbal agents within 14 days prior to initiation of study intervention:

<!-- -->

1. Known to be moderate or strong inhibitors or inducers of CYP3A4 (Appendix 9).
2. Known to be sensitive or narrow therapeutic index substrates of CYP3A4, CYP2C8, CYP2C9, or CYP2C19 (Appendix 10).

   - Prior treatment with any immunotherapy agent, including CD137 agonists or immune checkpoint blockade therapies (such as anti-cytotoxic T-lymphocyte-associated antigen-4 [anti-CTLA-4], anti-PD-1, and anti-PD-L1 therapeutic antibodies) and has experienced disease progression.
   * Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor agents) within two weeks prior to initiation of study intervention, or anticipation of need for systemic immunosuppressive medication during study intervention.

   NOTE: Participants who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Medical Monitor approval has been obtained.

   - Inadequately controlled arterial hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg), based on an average of three blood pressure readings on two sessions.

   NOTE: Anti-hypertensive therapy to achieve these parameters is allowable.

   - Prior history of hypertensive crisis or hypertensive encephalopathy.

   - Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within six months prior to initiation of study intervention.

   - History of hemoptysis (>2.5 mL of bright red blood per episode) within one month prior to initiation of study intervention.

   - Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).

   - Current or recent (within ten days of first dose of study intervention) use of aspirin (>325 mg/day) or treatment with dipyridamole, ticlopidine, clopidogrel, and cilostazol.

   - Current or recent (within ten days prior to initiation of study intervention) use of full dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose.

   NOTE: Allowable direct oral anticoagulants for prophylaxis include apixaban, edoxaban, rivaroxaban, and dabigatran. Participants should not be on any other anticoagulant for prophylaxis. Participants taking vitamin K antagonists, such as warfarin, are not eligible for the study.

   - Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within three days prior to the first dose of study intervention.

   - History of abdominal or tracheoesophageal fistula, GI perforation, or intra-abdominal abscess within six months prior to initiation of study intervention.

   - History of intestinal obstruction and/or clinical signs or symptoms of GI obstruction including sub-occlusive disease-related to the underlying disease or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding within six months prior to initiation of study intervention.

   NOTE: Participants with signs/symptoms of sub-/occlusive syndrome/intestinal obstruction at time of initial diagnosis may be enrolled if they had received definitive (surgical) treatment for symptom resolution.

   - Evidence of abdominal free air that is not explained by paracentesis or recent surgical procedure.
   * Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture.
   * Metastatic disease that involves major airways or blood vessels or centrally located mediastinal tumor masses (<30 mm from the carina) of large volume.
   * History of intra-abdominal inflammatory process within 6 months prior to initiation of study intervention, including but not limited to peptic ulcer disease, diverticulitis, or colitis.
   * Curative radiotherapy within 28 days and abdominal/pelvic radiotherapy within 60 days prior to initiation of study intervention, except palliative radiotherapy to bone lesions within seven days prior to initiation of study intervention.
   * Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to initiation of study intervention, or abdominal surgery, abdominal interventions or significant abdominal traumatic injury within 60 days prior to initiation of study intervention or anticipation of need for major surgical procedure during the course of the study or non-recovery from side effects of any such procedure.
   * Chronic daily treatment with a non-steroidal anti-inflammatory drug (NSAID). NOTE: Occasional use of NSAIDs for the symptomatic relief of medical conditions such as headache or fever is allowed. If the Investigator has specific considerations regarding the use of NSAIDs for pain management, it should be discussed with the Sponsor on a case-by-case basis.
   * Participant cannot swallow oral medications or have a GI illness that may clinically significantly affect the absorption of ABT-301 (e.g., chronic diarrhea with malabsorption).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Part I - To evaluate the safety and tolerability of escalating doses of ABT-301 in combination with fixed doses of tislelizumab 200 mg IV infusion and bevacizumab 7.5 mg/kg IV infusion Q3W, in participants with pMMR/non-MSI-H CRC. | From screening to 90 days after last dose
  Endpoints include:
  Adverse Event will be graded using the NCI CTCAE V5.0.
Part I - To determine the Maximum tolerated dose (MTD) and select the recommended Phase 2 dose (RP2D) of ABT-301. | From the first dose of ABT-301 to the completion of the first 21-day cycle of ABT-301 treatment in the last cohort.
  Endpoints include:
  Incidence of DLTs during the first cycle of treatment.
Part II - To evaluate the efficacy of two dosages/schemes of ABT-301 in combination with tislelizumab and bevacizumab. | From baseline until progression of disease or death, whichever occurs first. (up to 28 months)
  Endpoint:
  ORR per Investigator assessment, according to RECIST version 1.1.

SECONDARY OUTCOMES:
Part I - Objective Response Rate (ORR) per Investigator Assessment According to RECIST v1.1 | From baseline until progression of disease or death, whichever occurs first. (up to 28 months)
Part I - Duration of Response (DOR) per Investigator Assessment According to RECIST v1.1 | From baseline until progression of disease or death, whichever occurs first. (up to 28 months)
Part I - Progression-Free Survival (PFS) per Investigator Assessment According to RECIST v1.1 | From baseline until progression of disease or death, whichever occurs first. (up to 28 months)
Part I - Overall Survival (OS) | From baseline until progression of disease or death, whichever occurs first. (up to 28 months)
Part I - To characterize the PK of repeated doses of ABT-301 in participants with pMMR/non-MSI-H CRC. | From Cycle 1 Day 1 through Cycle 2 Day 1 (each cycle is 21 days)
  Maximum Plasma Concentration (Cmax) of ABT-301
Part I - To characterize the PK of repeated doses of ABT-301 in participants with pMMR/non-MSI-H CRC. | From Cycle 1 Day 1 through Cycle 2 Day 1 (each cycle is 21 days)
  Time to Reach Maximum Plasma Concentration (Tmax) of ABT-301
Part I - To characterize the PK of repeated doses of ABT-301 in participants with pMMR/non-MSI-H CRC. | From Cycle 1 Day 1 through Cycle 2 Day 1 (each cycle is 21 days)
  Area under the plasma concentration time curve from time zero to the time of the last quantifiable concentration (AUC₀-last) of ABT-301
Part I - To characterize the PK of repeated doses of ABT-301 in participants with pMMR/non-MSI-H CRC. | From Cycle 1 Day 1 through Cycle 2 Day 1 (each cycle is 21 days)
  Area Under the Plasma Concentration-Time Curve Over the Dosing Interval (AUC₀-τ) of ABT-301
Part I - To characterize the PK of repeated doses of ABT-301 in participants with pMMR/non-MSI-H CRC. | From Cycle 1 Day 1 through Cycle 2 Day 1 (each cycle is 21 days)
  Terminal Half-Life (t½) of ABT-301
Part I - To characterize the PK of repeated doses of ABT-301 in participants with pMMR/non-MSI-H CRC. | From Cycle 1 Day 1 through Cycle 2 Day 1 (each cycle is 21 days)
  Apparent Clearance (CL/F) of ABT-301
Part I - To characterize the PK of repeated doses of ABT-301 in participants with pMMR/non-MSI-H CRC. | From Cycle 1 Day 1 through Cycle 2 Day 1 (each cycle is 21 days)
  Apparent Volume of Distribution (Vz/F) of ABT-301
Part II - To evaluate the safety and tolerability of ABT-301 in combination with tislelizumab and bevacizumab. | From screening to 90 days after last dose
  Endpoints include:
  Adverse Event will be graded using the NCI CTCAE V5.0.
Part II - Objective Response Rate (ORR) per Investigator Assessment According to RECIST v1.1 | From baseline until progression of disease or death, whichever occurs first. (up to 28 months)
Part II - Duration of Response (DOR) per Investigator Assessment According to RECIST v1.1 | From baseline until progression of disease or death, whichever occurs first. (up to 28 months)
Part II - Progression-Free Survival (PFS) per Investigator Assessment According to RECIST v1.1 | From baseline until disease progression or death, whichever occurs first. (up to 28 months)
Part II - Overall Survival (OS) | From baseline until disease progression or death, whichever occurs first. (up to 28 months)
Part II - To evaluate the PK of ABT-301 in steady state. | From Cycle 1 Day 1 through the last Cycle Day 2 (each cycle is 21 days)
  Trough plasma concentration of ABT-301 in steady state and through plasma concentration of ABT-301 at specified timepoints.
Part II - To evaluate the PD of ABT-301 in steady state. | From Cycle 1 Day 1 through the last Cycle Day 2 (each cycle is 21 days)
  Level of AcH3 in PBMCs before and after treatment.

CONTACTS AND LOCATIONS:
Locations (15):
- Australia (8):
  - Liverpool Cancer Therapy Centre, Liverpool, New South Wales
  - Macquarie University Hospital (MUH), Macquarie Park, New South Wales
  - Scientia Clinical Research, Randwick, New South Wales
  - Greenslopes Private Hospital - Cyril Gilbert Cancer Centre, Greenslopes, Queensland
  - The Queen Elizabeth Hospital (TQEH), Woodville South, South Australia
  - Monash University - Faculty of Medicine, Nursing and Health Sciences, Clayton, Victoria
  - Austin Health - Cancer Clinical Trials Centre (CCTC), Heidelberg, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- Taiwan (7):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da Cancer Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital - Cancer Center, Taipei
  - Chang Gung Medical Foundation, Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided